CLINICAL TRIAL: NCT04303013
Title: A Randomized Controlled Trial of Guided Mindfulness Intervention During Radiotherapy.
Brief Title: Guided Meditation During Radiotherapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kimberly S. Corbin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-004546; NCI-2021-02757 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2020-02-26; First posted 2020-03-10 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-08

CONDITIONS: Quality of Life; Relaxation During Radiation Therapy; Cancer; Radiation Toxicity
MeSH Terms: conditions — Neoplasms; Radiation Injuries | interventions — Meditation; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care
- Meditation (Experimental)
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — Patients will attend weekly in person guided meditation sessions during the course of their radiation treatment. Patient will complete quality of life surveys before, during and after treatment.
  Arms: Meditation
Other: Standard of Care — Patient not assigned to meditation will undergo radiation with usual care and complete quality of life surveys before, during and after treatment.
  Arms: Standard of Care

SUMMARY:
The purpose of this research is to gather information on the effects of Mindfulness-Based Intervention (MBI) on quality of life during and after radiation treatment.

This study involves randomization. There is a 50 percent chance (like a flip of the coin) that you will be randomized to attend meditation sessions during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Prescribed a course of at least 15 daily fractions of RT for curative intent of any malignancy
* Willing to attend MBI sessions weekly during RT
* Able to transport themselves to scheduled MBI sessions in the DAHLC
* Able to complete questionnaire(s) by themselves
* Native English speaker (MBI sessions, videos, and QOL questionnaires are only available in English)
* ECOG Performance Status 0-2

Exclusion Criteria:

* Prescribed a course of RT with fewer than 15 consecutive, daily fractions
* Unable or unwilling to attend required MBI sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Meditation Sessions | Before radiation treatment.
  including emotional, physical, functional, and social domains assessed via the FACT-G during and after radiotherapy for the treatment of cancer.
Effectiveness of Meditation Sessions | During radiation treatment
  Comparison of change in total LASA-6 and single question relaxation surveys.
Effectiveness of Meditation Sessions | 3 months and 12 months post radiation treatment.
  Comparison of change in FACT-G, Promis 10 and LASA-6 surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly S. Corbin, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States